CLINICAL TRIAL: NCT02205723
Title: Smartphone-facilitated Medication Notification for Asthma Control in Pediatric Patients (SNAPP) Pilot Study
Brief Title: Smartphone-facilitated Asthma Control
Acronym: SNAPP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not initiated because we could not secure funding.
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Aerocrine AB (Industry)
Responsible Party: Principal Investigator, Donald H Arnold, Associate Professor of Pediatrics and Emergency Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB 140934
Record Dates: First submitted 2014-07-28; First posted 2014-07-31 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Childhood Asthma
Keywords: Asthma; Asthma exacerbations; Pediatric
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone Asthma Control (Experimental): Smartphone Asthma Control
  Interventions: Behavioral: Asthma teaching in ER; Behavioral: Smartphone Asthma Control
- Control (Active Comparator): Control group
  Interventions: Behavioral: Asthma teaching in ER

INTERVENTIONS:
Behavioral: Asthma teaching in ER — Asthma teaching
  Other Names: Asthma teaching
Behavioral: Smartphone Asthma Control — Smartphone Asthma Control
  Other Names: SNAPP
  Arms: Smartphone Asthma Control

SUMMARY:
The objective of this protocol is to pilot an innovative approach to medication adherence to determine if such an approach will improve inhaled corticosteroid (ICS) medication adherence, a critical gap in improving the health of children with asthma. SNAPP incorporates monitoring, reminders, and dynamic feedback through a smartphone that will improve ICS medication adherence and that the investigators believe will influence the child's future independence and chronic disease-management skills.

DETAILED DESCRIPTION:
The objective of this protocol is to pilot an innovative approach to medication adherence to determine if such an approach will improve inhaled corticosteroid (ICS) medication adherence, a critical gap in improving the health of children with asthma.

Acute asthma exacerbations occur yearly in almost 60% of children with asthma. They are the most frequent reason for childhood hospitalization and the most expensive component of pediatric asthma care in the U.S. Exacerbations impair quality of life and disproportionately affect African-American children, children with Medicaid insurance, and the poor. Up to 70% of exacerbations are preventable if guideline-recommended inhaled corticosteroid (ICS) medication adherence is achieved. However, ICS medication adherence in children with persistent asthma is dismal at only 11 - 18%. Amongst children with Medicaid insurance prescribed ICS, 63% discontinue the medication within 90 days. As a healthcare system, investigators have been unable to meaningfully improve ICS medication adherence in a cost-efficient way for patients with asthma, and particularly for the high-risk, highest-potential population of children with moderate or severe persistent asthma. These children suffer the greatest morbidity and mortality from asthma yet have highest-potential to benefit from improved ICS medication adherence. There is an urgent need for an efficacious adherence intervention for this population because, without it, these children will continue to experience impaired health and disproportionate morbidity.

The investigators' long-term objective is to identify and disseminate an intervention that will minimize the occurrence and severity of exacerbations in this population. The overall objective of this pilot study is to test the feasibility of Smartphone-facilitated medication Notification for Asthma Control in Pediatric Patients (SNAPP) using a wireless medication monitor (WMM) and smartphone application that provides parents reminders for administration of ICS medication, real-time feedback on preventive and controller medication adherence, and wireless upload of this data to a secure online database. The central hypothesis is that for children in this population, SNAPP will result in >=25% improved Asthma Control Test (ACT) scores in comparison with usual management. Secondary hypotheses are that the intervention will result in a >= 30% decrease in FeNO in comparison with usual care at 6 months and >=40% increase in ICS medication adherence at 6 months. The central hypothesis has been formulated on the basis of reports that parents of children with acute exacerbations continue to have insufficient knowledge of asthma self-management yet are motivated to do what is best for their child. SNAPP incorporates monitoring, reminders, and dynamic feedback through a smartphone that will improve ICS medication adherence and that will influence the child's future independence and chronic disease-management skills. Importantly, the investigators will use wireless medication monitors to accurately and objectively ascertain ICS medication adherence without patient effort. Parents are facile with and use wireless technology to organize their daily activities and for communicating. Incorporating this technology into health care and medication adherence is a logical next-step.

The investigators propose to test the hypotheses through the following Aim: To determine whether SNAPP meaningfully improves 6-month asthma control measured with the Asthma Control Test, airway inflammation measured using exhaled nitric oxide and ICS adherence compared with usual care, in an RCT of children with moderate or severe persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

1. TennCare Medicaid insurance, and an acute exacerbation (45% of our ED patients with acute asthma, section C.11.)
2. Parent has a smartphone and wireless account that they agree to use for this study (if randomized to intervention group), anticipated residence in the Nashville Metropolitan Service Area for at least 12 months, willingness to participate in phone-based (wireless or landline) ACT-scoring monthly, and willingness to return at 3, 6 and 12 months for FeNO testing.
3. The participant's PCP agrees that patient has moderate or severe persistent asthma and should be on ICS for at least the subsequent 12 months in accordance with NIH-NAEPP expert panel guidelines.87,88

Exclusion Criteria:

* Exclusion criteria include prior study enrollment, other medical condition contributing to respiratory distress (e.g., pneumonia, cystic fibrosis) or other diseases that may necessitate treatment with systemic corticosteroid (CCS; e.g., nephrotic syndrome).

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-12-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Childhood asthma control test | 6 months
  Measurement of change of C-ACT at 6 months.

SECONDARY OUTCOMES:
Fractional excretion of exhaled nitric oxide | 6 months
  Measurement of change of FeNO at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Donald H Arnold, MD, MPH, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt Children's Hospital, Nashville, Tennessee, United States